CLINICAL TRIAL: NCT07012031
Title: A Phase I/II Study Evaluating the Safety, Tolerability, and Efficacy of Sotorasib Plus Trastuzumab Deruxtecan in Patients With Advanced Non-Small Cell Lung Cancer With a KRASG12C Mutation
Brief Title: Sotorasib in Combination With Trastuzumab Deruxtecan for the Treatment of Locally Advanced and Metastatic Non-small Cell Lung Cancer With a KRAS G12C Mutation
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2025-03809; NCI-2025-03809 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MCC 23419; 10660 (Other: University Health Network Princess Margaret Cancer Center LAO); 10660 (Other: CTEP); UM1CA186644 (NIH)
Record Dates: First submitted 2025-05-29; First posted 2025-06-10 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Locally Advanced Lung Non-Small Cell Carcinoma; Metastatic Lung Non-Small Cell Carcinoma; Stage III Lung Cancer AJCC v8; Stage IV Lung Cancer AJCC v8
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Biopsy; Specimen Handling; Magnetic Resonance Spectroscopy; sotorasib; trastuzumab deruxtecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (trastuzumab deruxtecan, sotorasib) (Experimental): Patients receive trastuzumab deruxtecan IV over 30-90 minutes on day 1 and sotorasib PO QD on days 1-21 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients also undergo tumor biopsy and brain MRI at screening and ECHO or MUGA, CT, MRI and blood sample collection throughout the study. Additionally, patients with brain metastasis undergo brain MRI throughout the study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Echocardiography Test; Procedure: Magnetic Resonance Imaging; Procedure: Multigated Acquisition Scan; Drug: Sotorasib; Biological: Trastuzumab Deruxtecan

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo tumor biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNV Scan; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
Drug: Sotorasib — Given PO
  Other Names: AMG 510; AMG-510; AMG510; Lumakras; Lumykras
Biological: Trastuzumab Deruxtecan — Given IV
  Other Names: DS-8201; DS-8201a; Enhertu; Fam-trastuzumab Deruxtecan-nxki; T-DXd; WHO 10516

SUMMARY:
This phase I/II trial tests the safety, side effects and best dose of sotorasib with trastuzumab deruxtecan and how well the combination works in treating patients with KRAS G12C mutated non-small cell lung cancer that has spread to nearby tissues or lymph nodes (locally advanced) or that has spread from where it first started (primary site) to other places in the body (metastatic). Sotorasib blocks a protein made by the mutated KRAS gene (KRAS p.G12C), which may help keep tumor cells from growing and may kill them. It is a type of targeted therapy. Trastuzumab deruxtecan is in a class of medications called antibody-drug conjugates. It is composed of a monoclonal antibody, called trastuzumab, linked to a chemotherapy drug, called deruxtecan. Trastuzumab attaches to HER2 positive tumor cells in a targeted way and delivers deruxtecan to kill them. Giving sotorasib in combination with trastuzumab deruxtecan may be safe, tolerable, and/or effective in treating patients with locally advanced or metastatic non-small cell lung cancer with a KRAS G12C mutation.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety and tolerability of sotorasib (AMG-510) combined with trastuzumab deruxtecan (DS-8201a) in patients with advanced/metastatic non-small cell lung cancer (NSCLC) harboring a KRAS^G12C mutation who progress on a KRAS^G12C inhibitor and platinum-based chemotherapy with or without programmed cell death protein 1 (PD1)/programmed death-ligand 1 (PD-L1) inhibitors or PD1/L1 inhibitors alone. (Phase I) II. To determine overall response rate (ORR) defined as the proportion of patients with a confirmed response as per investigator assessment according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. (Phase II)

SECONDARY OBJECTIVES:

I. To observe and record anti-tumor activity. (Phase I) II. To determine the maximum tolerated dose (MTD) and the recommended phase II dose (RP2D) of trastuzumab deruxtecan (DS-8201a) and sotorasib (AMG-510) when combined. (Phase I) III. To estimate overall response rate (ORR) defined as the proportion of patients with a confirmed response as per investigator assessment according to RECIST version 1.1. (Phase I) IV. To estimate progression free survival (PFS). (Phase II) V. To estimate duration of response (DOR). (Phase II) VI. To estimate overall survival (OS). (Phase II) VII. To estimate adverse events (AEs) associated with the combination treatment. (Phase II)

EXPLORATORY OBJECTIVES:

I. To assess the rate of overexpression of ERBB2/ERBB3 gene expression by ribonucleic acid (RNA) sequencing (RNAseq) on NSCLC biopsy specimens collected at the pre-treatment timepoint in patients receiving sotorasib (AMG-510) + trastuzumab deruxtecan (DS-8201a). (Phase II) II. To estimate the correlation of ERBB2 gene expression measured by RNAseq on pre-treatment biopsies with response to the combination therapy and duration of response. (Phase II) III. To evaluate the pharmacokinetics (PK) of trastuzumab deruxtecan (DS-8201a) and sotorasib (AMG-510) and the immunogenicity of trastuzumab deruxtecan (DS-8201a). (Phase II)

OUTLINE: This is a phase I dose-escalation study of sotorasib in combination with trastuzumab deruxtecan (DS-8201a) followed by a phase II dose-expansion study.

Patients receive trastuzumab deruxtecan intravenously (IV) over 30-90 minutes on day 1 and sotorasib orally (PO) once daily (QD) on days 1-21 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients also undergo tumor biopsy and brain magnetic resonance imaging (MRI) at screening and echocardiography (ECHO) or multigated acquisition scan (MUGA), computed tomography (CT), MRI and blood sample collection throughout the study. Additionally, patients with brain metastasis undergo brain MRI throughout the study.

After completion of study treatment, patients are followed every 3 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically documented locally advanced or metastatic KRAS^G12C-mutant NSCLC that has previously been treated with a KRAS^G12C inhibitor AND an immune checkpoint inhibitor (ICI) AND chemotherapy, either given concurrently or sequentially, UNLESS they have any contra-indications to any drug class described above
* Patients must have KRAS^G12C mutation identified by tumor tissue or plasma circulating tumor deoxyribonucleic acid (ctDNA) profiling using a Clinical Laboratory Improvement Act (CLIA) certified College of American Pathologists (CAP) accredited platform; local molecular testing will be allowed. Testing must have been done within the last 5 years before enrollment in this study
* Data must be available for which prior KRAS^G12C inhibitor treatment the patient has received and the dates that they received it (type of KRAS^G12C inhibitor used and start and end dates must be collected prior to enrollment)
* Data must be available on the date patients received the last dose of KRAS^G12C inhibitor and the date of disease progression on their last treatment prior to screening for this trial. Data must be available on the last treatment they received and if it was not or did not include a KRAS^G12C inhibitor. The time between last KRAS^G12C inhibitor and treatment on this trial will be collected prior to enrollment
* Data must be available on historical HER2 immunohistochemistry (IHC) status (date of test, type of antibody used for the IHC test, scoring system [i.e., breast versus (vs.) gastric], and results must be collected prior to enrollment). Patients must also have ERBB2 (HER2) mutations status identified by tumor tissue or plasma ctDNA profiling; local (i.e., commercial or institutional next generation sequencing [NGS]) molecular testing will be allowed. Patients who do not have this information available for collection will not be enrolled on this study
* Patients must have measurable disease, as defined by RECIST v1.1 using computed tomography (CT) or magnetic resonance imaging (MRI). Previously irradiated lesions cannot be counted as target lesions unless there has been demonstrated progression in the lesions since radiotherapy and no other lesions are available for selection as target lesions
* Age ≥ 18 years at date of informed consent form signature

  * Because no dosing or adverse event data are currently available on the use of sotorasib (AMG-510) in combination with trastuzumab deruxtecan (DS-8201a) in patients < 18 years of age, children are excluded from this study
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 (Karnofsky ≥ 60%)
* Hemoglobin ≥ 9 g/dL (within 14 days of enrollment)
* Leukocytes ≥ 3,000/mcL (within 14 days of enrollment)
* Absolute neutrophil count ≥ 1,500/mcL (within 14 days of enrollment)

  * No administration of granulocyte colony stimulating factor (G-CSF) is allowed within 1 week prior to screening assessment
* Platelets ≥ 100,000/mcL (within 14 days of enrollment)

  * No transfusions with red blood cells or platelets are allowed within 1 week prior to screening assessment
* Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN) (within 14 days of enrollment), (< 3 x ULN in the presence of documented Gilbert's syndrome or liver metastases at baseline)
* Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT)(serum glutamic pyruvic transaminase [SGPT]) ≤ 3 x institutional ULN (within 14 days of enrollment) (< 5 x ULN in participants with liver metastases)
* Serum albumin ≥ 2.5 g/dL (within 14 days of enrollment)
* International normalized ratio (INR)/prothrombin time (PT) and activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN (within 14 days of enrollment)
* Creatinine ≤ 1.5 x institutional ULN OR creatinine clearance (CrCL) ≥ 30 mL/min/ as determined by (using actual body weight) (within 14 days of enrollment)
* Patients must have left ventricular ejection fraction (LVEF) ≥ 50% by either an echocardiogram (ECHO) or multigated acquisition (MUGA) scan within 28 days before enrollment
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients with treated brain metastases are eligible with 1 day washout for stereotactic radiosurgery (SRS) and 2 weeks washout for whole brain radiation (WBRT)
* Patients with new or progressive brain metastases (active brain metastases) are eligible if the treating physician determines that immediate central nervous system (CNS) specific treatment is not required and is unlikely to be required during the first cycle of therapy
* Patients must have a life expectancy of ≥ 12 weeks
* Patients must have a corrected QT interval (QTc) ≤ 470 msec for women and ≤ 450 msec for men (based on average screening triplicates)
* Patients must be willing to undergo a mandatory pre-treatment biopsy (28 days before treatment starts on cycle 1 day 1 [C1D1]) for patients enrolled into the expansion phase (phase II). The pre-treatment biopsy is optional for patients enrolled into the dose escalation phase (phase I)
* Patients must have the ability to ingest and retain oral (PO) medications
* The effects of the combination of sotorasib (AMG-510) and trastuzumab deruxtecan (DS-8201a) on the developing human fetus are unknown. For this reason and because HER-2-directed antibody conjugated to a topoisomerase 1 inhibitor agents are known to be teratogenic, women of child-bearing potential (WOCBP) must agree to use dual methods of contraception and must have a negative serum pregnancy testing at screening. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Women treated or enrolled on this protocol must agree to use a highly effective method of contraception, if sexually active, or avoid intercourse during the study treatment and for 7 months following the last dose of study drug. Sotorasib (AMG-510) may reduce the effectiveness of hormonal contraceptives, and therefore women using hormonal contraceptives should add a barrier method on study and for an additional 7 days after the last dose of sotorasib (AMG-510). Men treated or enrolled on this protocol must also agree to use a highly effective barrier method of contraception, if sexually active, or avoid intercourse throughout the duration of the study and for 4 months following the last dose of study drug. To prevent exposure of the unborn child to sotorasib (AMG-510) through semen, male subjects will be required to practice true sexual abstinence (not have sex) or must wear a condom during vaginal sex
* Women of non-child-bearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea (in questionable cases, a blood sample with simultaneous follicle-stimulating hormone [FSH] > 40 mIU/mL and estradiol < 40 pg/mL [< 147 pmol/L] is confirmatory) are eligible. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods outlined for women of child-bearing potential if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment. For most forms of HRT, at least 2-4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method
* Male subjects must not freeze or donate sperm starting at screening and throughout the study period, and at least 4 months after the final study drug administration. Preservation of sperm should be considered prior to enrollment in this study
* Female subjects must not donate, or retrieve for their own use, ova from the time of screening and throughout the study treatment period, and for at least 7 months after the final study drug administration
* Ability to understand and the willingness to sign a written informed consent document. Legally authorized representatives may sign and give informed consent on behalf of study participants

Exclusion Criteria:

* Patients with a history of (non-infectious) interstitial lung disease (ILD) that required steroids, has current ILD, or where suspected ILD cannot be ruled out by imaging at screening. These patients will be excluded because trastuzumab deruxtecan (DS-8201a) is known to increase the risk of developing ILD and pneumonitis
* Patients with clinically severe pulmonary compromise resulting from intercurrent pulmonary illnesses including, but not limited to, any underlying pulmonary disorder (i.e., pulmonary emboli within three months of the study enrollment, severe asthma, severe chronic obstructive pulmonary disease [COPD], restrictive lung disease, prior complete pneumonectomy), and any autoimmune, connective tissue or inflammatory disorders (e.g., rheumatoid arthritis, Sjogren's, sarcoidosis, etc.) where there is documented or a suspicion of pulmonary involvement or pneumonectomy at the time of screening. These patients will be excluded because trastuzumab deruxtecan (DS-8201a) is known to increase the risk of developing ILD and pneumonitis
* Patients who have had chest radiation therapy within 4 weeks (2 weeks for palliative stereotactic body radiation therapy). These patients will be excluded because trastuzumab deruxtecan (DS-8201a) and sotorasib (AMG-510) are known to increase the risk of developing pneumonitis
* Patients who have had a major surgery and are not yet fully healed from surgical incisions
* Patients who have had prior treatment with an antibody drug conjugate with a topoisomerase 1 inhibitor payload (i.e., sacituzumab govitecan, datopotomab deruxtecan, or trastuzumab deruxtecan) or with a topoisomerase inhibitor
* Patients with a history of significant lung disease requiring systemic corticosteroids treatment (> 10 mg of prednisone daily) within the last six months of registration
* Based on pre-clinical data, trastuzumab deruxtecan (DS-8201a) is associated with corneal disease. Patients with clinically significant corneal disease, in the opinion of the investigator, will be excluded from this study
* Patients with spinal cord compression, defined as untreated and symptomatic, or requiring therapy with corticosteroids or anticonvulsants to control associated symptoms
* Patients with an uncontrolled infection requiring IV antibiotics, antivirals, or antifungals
* Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > grade 1) with the exception of alopecia. Subjects with chronic grade 2 toxicities (i.e., defined as no worsening to > grade 2 for at least 3 months prior to first exposure to study intervention and managed with standard of care treatment) may be eligible per the discretion of the investigator after consultation with the sponsor medical monitor or designee (e.g., grade 2 chemotherapy-induced neuropathy). Subjects should no longer be symptomatic nor require treatment with corticosteroids (prednisone > 10 mg or equivalent) or anticonvulsants and must have recovered from the acute toxic effect of radiotherapy
* Patients who are receiving any other investigational agents
* Patients with a history of allergic reactions attributed to compounds of similar chemical or biologic composition to sotorasib (AMG-510), such as adagrasib, or trastuzumab deruxtecan (DS-8201a)
* Patients who have a history of severe hypersensitivity reactions to other monoclonal antibodies
* Patients who are taking strong CYP3A4 inducers should be switched to an alternative drug
* Avoid coadministration with P-glycoprotein (P-gp) substrates for which minimal concentration changes may lead to serious toxicities. If coadministration cannot be avoided, dose adjustment of the substrate may be required. Please refer to the prescribing information for the substrate
* Patients with uncontrolled intercurrent illness or any other significant condition(s) that would make participation in this protocol unreasonably hazardous or interfere with the evaluation of the clinical study results
* Pregnant women are excluded from this study because trastuzumab deruxtecan (DS-8201a) is a HER2-directed antibody conjugated to a topoisomerase 1 inhibitor agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with trastuzumab deruxtecan (DS-8201a) breastfeeding should be discontinued if the mother is treated with trastuzumab deruxtecan (DS-8201a). These potential risks may also apply to other agents used in this study
* Patients with uncontrolled or significant cardiovascular disease (i.e., history of myocardial infarction within 6 months from screening, symptomatic congestive heart failure [CHF] [New York Heart Association class II to IV], troponin levels consistent with myocardial infarction 28 days prior to enrollment, history of unstable angina, or serious cardiac arrhythmia)
* Patients with prior history of pneumonitis grade 2 or higher or ILD
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patients unable to receive both iodinated contrast for CT scans and gadolinium contrast for MRI scans
* Patients that have pleural effusion, ascites, or pericardial effusion that requires drainage within 2 weeks of study screening procedures, peritoneal shunt, or cell-free and concentrated ascites reinfusion therapy (CART)
* Patients that have received a live vaccine within 30 days prior to the first dose of study drug will be excluded. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, bacillus Calmette- Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2026-08-07 (Estimated); Primary Completion 2027-06-14 (Estimated); Study Completion 2027-06-14 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicities of combined trastuzumab deruxtecan (DS-8201a) and sotorasib (AMG-510) treatment (Phase I) | Within the first 21 days of treatment initiation
  Will be defined as an adverse event (AE) that is at least possibly related to the study treatment. Severity will be graded according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0.
Overall response rate (ORR) (Phase II) | Up to 5 years
  Will be defined as the proportion of patients with a confirmed response as per investigator assessment according to Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1. Will be plotted using Kaplan-Meier method.

SECONDARY OUTCOMES:
Maximum tolerated dose (MTD)/recommended phase 2 dose (RP2D) of trastuzumab deruxtecan (DS-8201a) and sotorasib (AMG-510) combination (Phase I) | Up to 5 years
  Will be determined based on the totality of safety, tolerability, and clinical activity data as appropriate. RP2D nay be determined to be the highest dose level, the MTD, or it may be a lower dose based on the consensus of the investigators, Cancer Therapy Evaluation Program, and pharmaceutical company collaborators.
ORR (Phase I) | Up to 5 years
  Will be defined as the proportion of patients with a confirmed response (i.e., response confirmed by a second radiographic evaluation) as per investigator assessment according to RECIST v 1.1. Will be summarized using both a point estimate and its exact 95% confidence interval based on the binomial distribution.
Progression-free survival (PFS) (Phase II) | From start of treatment to disease progression or death due to any cause, assessed up to 5 years
  Will be plotted using Kaplan-Meier method.
Duration of response (Phase II) | From the time measurement criteria are first met for complete response or partial response until the first date that recurrent or progressive disease is objectively documented, assessed up to 5 years
  Will be plotted using Kaplan-Meier method.
Overall survival (OS) (Phase II) | From first treatment to time of death due to any cause, assessed up to 5 years
  Will be plotted using Kaplan-Meier method.
Incidence of AEs (Phase II) | Up to 30 days after the last dose of study drug
  Will be tabulated by grade. AEs will be described and graded using NCI CTCAE v 5.0.
Rate of ERBB2/ERBB3 gene overexpression (Phase II) | At pre-treatment
  Gene expression levels will be measured by counts (i.e., by the number of reads mapped on each gene). Data analysis will be descriptive statistics in nature (e.g., proportion of ERBB2/ERBB3 gene expression in each response group).
Correlation between ERBB2 gene expression in pre-treatment specimens and the treatment response (Phase II) | Up to 5 years
  Will be measured by ribonucleic acid (RNA)-Sequencing.

OTHER OUTCOMES:
Correlation between HER2 immunohistochemistry (IHC) archival and pre-treatment (study biopsy) results and ORR, PFS, and OS (Phase II) | Up to 5 years
  Data analysis will be descriptive statistics in nature (e.g., proportion of IHC+ or proportion of overexpressed in each response group).
Correlation between ERBB2 gene expression and ORR, PFS, and OS (Phase II) | Up to 5 years
  Will be measured by RNA Salah Targeted Expression Panel and mass spectrometry.
Correlation between circulating tumor deoxyribonucleic acid (ctDNA) clearance and ORR, PFS, and OS (Phase II) | Up to 5 years
  Kaplan Meier method will be used to estimate the median PFS and OS for the ctDNA clearance and non-clearance groups.
Whole exome sequencing (WES) (Phase II) | Up to 5 years
Correlation between WES and response rate, PFS, and OS (Phase II) | Up to 5 years
Pharmacokinetics of trastuzumab deruxtecan (DS-8201a) (Phase II) | Before trastuzumab deruxtecan (DS-8201a) infusion and within 30 minutes of the end of infusion on cycle (c) 1 day (d) 1, C2D1, C4D1, and C6D1
Pharmacokinetics of sotorasib (AMG-510) (Phase II) | Before sotorasib dose and trastuzumab deruxtecan (DS-8201a) infusion on C1D1, C2D1, C6D1 and within 30 minutes of the end of DS-8201a (T-DXd) infusion on C1D1 and C2D1
Antidrug antibodies against trastuzumab deruxtecan (DS-8201a) (Phase II) | Before trastuzumab deruxtecan (DS-8201a) infusion on C1D1, C2D1, C4D1, C6D1 and at the end of treatment visit

CONTACTS AND LOCATIONS:
Overall Officials: Andreas N Saltos, Principal Investigator — University Health Network Princess Margaret Cancer Center LAO
Locations (1):
- University Health Network Princess Margaret Cancer Center LAO, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm